CLINICAL TRIAL: NCT00711932
Title: Death Receptor-Mediated Apoptosis and Therapy Strategies in Ovarian Cancer
Brief Title: The Effect of TRA-8 on Ovarian Cancer Tissue
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tong Zhou, MD, Associate Professor of Medicine, University of Alabama at Birmingham
Other Study IDs: F080328006/UAB0802; ROI CA 123197-01
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; TRA-8; Monoclonal Antibody; Tissue Slice Technology
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to determine the apoptosis-inducing efficacy of TRA-8 in patient ovarian cancer tissues using a tissue slice technology. In addition, we want to evaluate the expression of apoptosis regulatory proteins using multiplex proteomic technology and its correlation with TRA-8-induced cytotoxicity in patient ovarian cancer tissues.

DETAILED DESCRIPTION:
Ovarian cancer remains highly lethal, with an estimated 25,580 new cases and 16,090 death per year in the US. The most common ovarian cancers arise from the surface epithelium of the ovary. Approximately 75% of patients with advanced-stage cancer are surgically incurable. While chemotherapy is a critical component of treatment, the pre-existing and induced chemoresistance of ovarian cancer cells is a major obstacle in treatment of patients with advanced disease. Novel strategies to enhance the established therapeutic Defective apoptosis has been proposed as one of the major mechanisms that lead to malignant transformation and resistance to therapeutics. Defective apoptosis may result from increased growth stimulation (oncogenes), decreased growth inhibition (tumor suppressor genes) or imbalanced apoptosis regulation. Alterations of the Bcl-2 family proteins have been reported to be associated with chemotherapy resistance in ovarian cancer cells.(1) Increased anti-apoptosis protein, Bcl-XL, may play a role in preventing apoptosis of ovarian cancer cells in response to chemotherapy. Conversely, high levels of pro-apoptosis protein, Bax, are associated with a favorable response to therapy. The role of these and other apoptotic regulatory proteins in sensitivity/resistance mechanisms to chemotherapy in patient's ovarian cancer cells are just beginning to be elucidated.

Precision cut tumor slices will be prepared from fresh primary ovarian tumor specimens using the Krumdieck tissue slicer, followed by ex vivo TRA-8 cytotoxicity assays on the tumor slices. Tumor-derived tissue slices may be used immediately in short term assays with no need to isolate or expand tumor cells, thus avoiding potential problems in maintaining cell viability or selecting variant cells during tumor dispersion or longer periods of in vitro cell culture. Demonstration of TRA-8-induced apoptosis using primary ovarian tumors in ex vivo tumor slice cytotoxicity assays can strengthen the rationale for this therapy in this tumor type and may be used to select patients who would most likely benefit from TRA-8 therapy. The sensitivity of ovarian patient tumors to TRA-8, paclitaxel, and carboplatin will be evaluated in tumor slice cytotoxicity assays as single agents and in combination. Slices from different treatment conditions will be paraffin-embedded or frozen for immunohistochemical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have suspected ovarian cancer and must be a candidate for surgery.
* Patients must have provided a signed consent form.
* Patients must have extra tumor at the time of surgery that is appropriate for tumor slicing.
* Patients must be at least 19 years of age.
* Patients must have histologically confirmed epithelial carcinoma of the ovary or of extra-ovarian origin, any histologic subtype or stage.

Exclusion Criteria:

* Patients who have received any prior therapy for ovarian cancer.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed epithelial carcinoma of the ovary or of extra-ovarian origin, any histologic subtype or stage 19 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Presence of TRA-8 apoptosis | At the time of surgery
  Apoptosis properties of TRA-8 will be analyzed in tissue collected from surgery using tissue slice technology.
Presence of apoptosis regulatory proteins | At the time of surgery
  The presence of apoptosis regulatory properties will be analyzed in tissue collected from surgery using multiplex proteomic technology.

CONTACTS AND LOCATIONS:
Overall Officials: Tong Zhou, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States